CLINICAL TRIAL: NCT06960317
Title: Expanding the Use of Paracervical Block for IUD Placements and Adding a Compassionate Care Assessment
Brief Title: Empathy Through Pain Control: Lidocaine Paracervical Block for IUD Placements
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 812390
Record Dates: First submitted 2025-04-16; First posted 2025-05-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Contraception; Pain, Acute; Anesthesia, Local
MeSH Terms: conditions — Acute Pain | interventions — phenylmercury borate

STUDY DESIGN:
Intervention Model Description: 6-armed single-blind randomized controlled
Who Masked: Participant
Masking Description: Participants will not know their group assignment. The clinicians will know which group the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 1a: Buffered lidocaine paracervical block (Experimental): Treatment group: will receive a 20-mL buffered (2 cc of sodium bicarbonate, 18 cc of 1% lidocaine) paracervical block administered before IUD placement. They will also receive 2 cc of buffered 1% lidocaine at the top of the cervix where the clinician places a tenaculum.
  Interventions: Drug: Buffered Lidocaine
- 1b: Capped needle (Sham Comparator): Sham group: will receive a capped needle without any medication administered as paracervical block before IUD placement. They will receive 2 cc of buffered 1% lidocaine at the top of the cervix where the clinician places a tenaculum.
  Interventions: Other: Sham Comparator
- 2a: Buffered lidocaine paracervical block (Experimental): Treatment group: will receive a 20-mL buffered (2 cc of sodium bicarbonate, 18 cc of 1% lidocaine) paracervical block administered before IUD placement. They will also receive 2 cc of buffered 1% lidocaine at the top of the cervix where the clinician places a tenaculum.
  Interventions: Drug: Buffered Lidocaine
- 2b: Unbuffered lidocaine paracervical block (Active Comparator): Active comparator group: will receive a 20-mL unbuffered (1% lidocaine) paracervical block administered before IUD placement. They will also receive 2 cc of buffered 1% lidocaine at the top of the cervix where the clinician places a tenaculum.
  Interventions: Drug: Unbuffered lidocaine
- 3a: Medicated gel (Experimental): Treatment group: will receive lidocaine-infused gel prior to administration of paracervical block.
  Interventions: Drug: Xylocaine jelly 2%
- 3b: Non-medicated gel (Placebo Comparator): Placebo group: will receive a non-medicated gel prior to administration of paracervical block.
  Interventions: Drug: Surgilube

INTERVENTIONS:
Drug: Buffered Lidocaine — To determine if a 20 cc buffered (2 cc of sodium bicarbonate, 18 cc of 1% lidocaine) lidocaine paracervical block decreases pain with IUD placement
  Arms: 1a: Buffered lidocaine paracervical block; 2a: Buffered lidocaine paracervical block
Other: Sham Comparator — None - capped needle will not be injected nor will it contain any medication.
  Arms: 1b: Capped needle
Drug: Unbuffered lidocaine — To determine if a 20 cc unbuffered (1% lidocaine) lidocaine paracervical block decreases pain with IUD placement
  Arms: 2b: Unbuffered lidocaine paracervical block
Drug: Xylocaine jelly 2% — To determine if a Xylocaine jelly (2% infused lidocaine) decreases pain with paracervical block
  Arms: 3a: Medicated gel
Drug: Surgilube — To determine if a placebo gel is inferior to lidocaine gel for pain with paracervical block
  Arms: 3b: Non-medicated gel

SUMMARY:
The goal of this research study is to learn more about how different uses of a numbing medication might affect pain levels while getting an IUD placed. The investigators are also studying participants opinions of their clinicians' empathy.

The investigators are inviting patients who arrive at their clinic visit seeking an IUD.

Usually, at University of California, San Diego (UCSD), for patients who have never delivered a baby, clinicians use a buffered paracervical block for before IUD placement. The purpose of this research study is to investigate whether a "buffered" (2 cc of sodium bicarbonate, 18 cc of 1% lidocaine) paracervical block (numbing medication given on both sides of the cervix) is effective in reducing pain during IUD placement in individuals with prior C-sections, the difference between buffered and unbuffered for nulliparous patients, and whether a medicated gel reduces pain with the paracervical block.

DETAILED DESCRIPTION:
Lidocaine is a drug that has been approved by the Food and Drug Administration (FDA). Sodium bicarbonate is an additive that buffers the acidity of lidocaine. The combination of the two is safe and effective as a paracervical block for pain relief in various OBGYN procedures. At UCSD and other places, it is not currently standard practice for people with prior deliveries birth to receive a paracervical block prior to IUD placement.

Participants who take part in this study, may receive an injection of buffered lidocaine (2 cc of sodium bicarbonate, 18 cc of 1% lidocaine), an injection of unbuffered block, and/or lidocaine gel.

Throughout the local anesthetic and intrauterine device (IUD) placement procedure, research team members will present participants with questionnaires to complete to assess participants' pain, participants' satisfaction with the procedure, and how much empathy participants feel the clinician has shown.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Women IUD placement for contraception or heavy menstrual bleeding
3. Ages 18-50
4. English-speaking
5. Participants must not have a past medical history of substance use disorders, pain disorders, use of prescription pain medications or are found to be pregnant

Exclusion Criteria:

1. No history of vaginal delivery
2. Current use of prescription pain medication prior to procedure. Over-the-counter medications such as those containing ibuprofen, aspirin, acetaminophen, or naproxen are allowed.
3. Diagnosed chronic pain condition
4. Current pregnancy
5. Known allergic reactions to components of the local anesthetic
6. History of an IUD placement
7. Current substance use or history of substance use
8. Known contraindications to IUD, such as unexplained vaginal bleeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain scores during IUD placement procedure | From speculum placement to 5 minutes post-procedure
  Does buffered 1% lidocaine paracervical block decrease pain during IUD. placement procedures. Pain will be measured on a 10-cm Visual Analog Scale (VAS) with score points ranging from 0-10, where 0 means "No pain" and 10 means "Worst pain possible."

SECONDARY OUTCOMES:
Patient perceptions of clinician empathy | From pre-procedure baseline to 5 minutes post-procedure
  What is the relationship between pain and feelings about clinician empathy. Empathy will be measured through answers to the 10-question Consultation and Relational Empathy (CARE) Measure. Each question is answered by a 5-point scale of how well the patient believes their clinician to be at various types of empathetic gestures, where 1 equals "poor" and 5 equals "excellent."

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K Mody, MD, MPH, Principal Investigator — UC San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin J, Kaneshiro B, Elia J, Raidoo S, Savala M, Soon R. Buffered lidocaine for paracervical blocks in first-trimester abortions: a randomized controlled trial. Contracept X. 2020 Oct 18;2:100044. doi: 10.1016/j.conx.2020.100044. eCollection 2020. PMID 33196038
- [Background] Azizkhani R, Forghani M, Maghami-Mehr A, Masomi B. The effects of injections of warmed bicarbonate-buffered Lidocaine as a painkiller for patients with trauma. J Inj Violence Res. 2015 Jul;7(2):87-8. doi: 10.5249/jivr.v7i2.523. Epub 2013 Dec 12. No abstract available. PMID 24879075
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Welch MN, Czyz CN, Kalwerisky K, Holck DE, Mihora LD. Double-blind, bilateral pain comparison with simultaneous injection of 2% lidocaine versus buffered 2% lidocaine for periocular anesthesia. Ophthalmology. 2012 Oct;119(10):2048-52. doi: 10.1016/j.ophtha.2012.05.029. Epub 2012 Jul 6. PMID 22771049
- [Background] Narvaez J, Wessels I, Bacon G, Chin VR, Baqai WK, Zimmerman GJ. Prospective randomized evaluation of short-term complications when using buffered or unbuffered lidocaine 1% with epinephrine for blepharoplasty surgery. Ophthalmic Plast Reconstr Surg. 2010 Jan-Feb;26(1):33-5. doi: 10.1097/IOP.0b013e3181b80c13. PMID 20090482
- [Background] Hobeich P, Simon S, Schneiderman E, He J. A prospective, randomized, double-blind comparison of the injection pain and anesthetic onset of 2% lidocaine with 1:100,000 epinephrine buffered with 5% and 10% sodium bicarbonate in maxillary infiltrations. J Endod. 2013 May;39(5):597-9. doi: 10.1016/j.joen.2013.01.008. Epub 2013 Mar 20. PMID 23611375
- [Background] Harreld TK, Fowler S, Drum M, Reader A, Nusstein J, Beck M. Efficacy of a Buffered 4% Lidocaine Formulation for Incision and Drainage: A Prospective, Randomized, Double-blind Study. J Endod. 2015 Oct;41(10):1583-8. doi: 10.1016/j.joen.2015.06.017. Epub 2015 Aug 4. PMID 26253800
- [Background] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115
- [Background] Allen RH, Raker C, Goyal V. Higher dose cervical 2% lidocaine gel for IUD insertion: a randomized controlled trial. Contraception. 2013 Dec;88(6):730-6. doi: 10.1016/j.contraception.2013.07.009. Epub 2013 Aug 1. PMID 24012096